CLINICAL TRIAL: NCT00392964
Title: Patterns of Antiacids Use in Patients With IHD Admitted to Department of Internal Medicine
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Other Study IDs: ZSA2438CTIL
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Ischemic Heart Disease
Keywords: Antacids; Proton pump inhibitors; aspirin; ischemic heart disease; Dyspepsia
MeSH Terms: conditions — Myocardial Ischemia; Dyspepsia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is substantial, continuing, and unexplained rise in prescribing of proton pump inhibitors. It is unknown whether their use in practice has corresponded to their licensed indications.

Although the indications for H2RA or PPI administration in the treatment of acid-related diseases and the prevention of gastric mucosal damage have been well defined in the medical literature, the perception of benefit from their use frequently tends to be extrapolated to all patients in general, leading to an excessive consumption of these drugs in general practice.

To date, however, little has been published with regard to the overall use or misuse of these drugs in hospital populations in ischemic heart disease patients as a secondary prevention to Aspirin use.

We will undertake a 6-months retrospective survey (about 1200 patients) to evaluate the use of acid-suppressive medications in the general internal medicine ward of Rambam Hospital.

We will extract all records of prescribing of a proton pump inhibitor within Rambam Hospital computerized patients file program (Premetheuos) in period of half year, categorized and analyze them using statistical X2 test.

DETAILED DESCRIPTION:
Dyspeptic symptoms are a common presenting complaint, and there is continuing debate about management. Acid suppressant drugs, the most potent of which are proton pump inhibitors, are often prescribed, and it has been suggested that proton pump inhibitors are probably too widely prescribed for minor symptoms, and the cost implications of this are clear. There is substantial, continuing, and unexplained rise in prescribing of proton pump inhibitors. It is unknown whether their use in practice has corresponded to their licensed indications.

Although the indications for H2RA or proton pump inhibitor administration in the treatment of acid-related diseases and the prevention of gastric mucosal damage have been well defined in the medical literature, the perception of benefit from their use frequently tends to be extrapolated to all patients in general, leading to an excessive consumption of these drugs in general practice.

In addition, Physicians, nowadays tend to prescribe proton pump inhibitors for cardiac patients who use aspirin as secondary prevention of their illness.

To date, however, little has been published with regard to the overall use or misuse of these drugs in hospital populations, or to the fall-out of hospital prescriptions in general practice and none has been published regarding its use in ischemic heart disease patients as a secondary prevention to Aspirin use.

We will undertake a 6-months retrospective survey (about 1200 patients) to evaluate the use of acid-suppressive medications in the general internal medicine ward of Rambam Hospital, a large teaching hospital in Northern Israel; as well as the appropriateness of their prescription to the licensed indications, while dividing them to subgroups of ischemic heart disease patients.

We will extract all records of prescribing of a proton pump inhibitor within Rambam Hospital computerized patients file program (Premetheuos) in period of half year, categorized and analyze them using statistical X2 test.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic Heart Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 2006-01; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zaher S Azzam, MD, Principal Investigator — Acting Director of Internal Medicine "B"
Locations (2):
- Israel (2):
  - Rambam: Health Care Campus, Haifa
  - Rambam Health Care Campus, Haifa